CLINICAL TRIAL: NCT07033260
Title: The Predictive Value of Carotid Corrected Flow Time and Peak Flow Velocity Variability for Intradialytic Hypotension: A Prospective Multicenter Observational Study
Brief Title: Predictive Value of Carotid Ultrasonography for Intradialytic Hypotension
Acronym: CUPID
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Wannan Medical College (Other)
Collaborators: Wuhu City Second People's Hospital (Other); Wuhu County Traditional Chinese Medicine Hospital (Other)
Responsible Party: Principal Investigator, Qiancheng Xu, Principal Investigator, First Affiliated Hospital of Wannan Medical College
Other Study IDs: 2025-12
Record Dates: First submitted 2025-06-14; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Intradialytic Hypotension; End-Stage Renal Disease Requiring Haemodialysis; Uremia; Chronic; Hemodialysis
Keywords: Carotid ultrasonography; Corrected flow time; Peak flow velocity variability; Intradialytic hypotension; Hemodialysis; Ultrasonographic predictors; Vascular ultrasonography; Fluid management; Dialysis safety
MeSH Terms: conditions — Uremia; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Maintenance Hemodialysis Patients: Adult patients aged 18 to 80 years undergoing maintenance hemodialysis for more than three months. All participants will undergo carotid ultrasonography to measure corrected flow time (FTc) and peak flow velocity variability (PFVV) during routine dialysis sessions. The study aims to evaluate the association between these ultrasonographic parameters and the occurrence of intradialytic hypotension.
  Interventions: Other: Non-invasive Monitoring

INTERVENTIONS:
Other: Non-invasive Monitoring — All participants will undergo non-invasive ultrasonographic measurement of carotid corrected flow time (FTc) and peak flow velocity variability (PFVV) before and during hemodialysis sessions. No treatment or experimental intervention will be applied.

SUMMARY:
This multicenter, prospective observational study aims to evaluate the predictive value of carotid corrected flow time (FTc) and peak flow velocity variability (PFVV) for hypotension during maintenance hemodialysis. Conducted at The First Affiliated Hospital of Wannan Medical College, Wuhu City Second People's Hospital, Wuhu Hospital of Chinese Traditional Medicine, Wuhu Jinghu District Hospital, and Wuhu Guangji Hospital, the study will include adult patients (≥18 years) with end-stage renal disease (ESRD) on long-term hemodialysis for at least three months. Patients with acute kidney injury, severe cardiac conditions, or other factors affecting results will be excluded. Ultrasound assessments of FTc and PFVV will be performed once, at 1 hour after dialysis initiation. Blood pressure will be monitored during the procedure. The primary outcome is to determine the sensitivity, specificity, and optimal cutoff points of FTc and PFVV in predicting intradialytic hypotension. The estimated sample size is 183 participants, with analysis performed using ROC curves and multivariate regression. The protocol complies with ethical standards and aims to develop a simple, non-invasive, real-time tool to improve patient safety and individualized management during hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18 to 80 years. Diagnosed with end-stage renal disease (ESRD). Undergoing maintenance hemodialysis for more than three months. Willing and able to provide informed consent and comply with study procedures.

Exclusion Criteria:

Patients with significant carotid artery stenosis due to heavy atherosclerotic plaque (defined as more than 70% stenosis confirmed by ultrasound or angiography).

Hemodynamically unstable patients or those requiring vasopressor support. Patients with significant arrhythmias (e.g., atrial fibrillation, ventricular tachycardia).

Dialysis sessions terminated for reasons unrelated to hypotension (e.g., technical issues, patient request).

Use of antihypertensive medications during dialysis sessions. Inability to undergo ultrasound assessment due to factors such as severe obesity or wounds obstructing access.

Patients who withdraw informed consent during the study.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18 to 80 years with end-stage renal disease who have been receiving maintenance hemodialysis for more than three months at participating dialysis centers. Participants are required to be able to provide informed consent and cooperate with study procedures.
Sampling Method: Non-Probability Sample
Enrollment: 183 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Predictive Value of Carotid Corrected Flow Time (FTc) for Intradialytic Hypotension | 1 hour after dialysis start during a single session.
  The carotid corrected flow time (FTc) is the duration of blood flow in the carotid artery, corrected for heart rate, measured using ultrasonography at 1 hour after hemodialysis initiation. This parameter will be evaluated for its ability to predict hypotension episodes during dialysis, with analysis focusing on sensitivity, specificity, and ROC curve to determine diagnostic accuracy.
Predictive Value of Peak Flow Velocity Variability (PFVV) for Intradialytic Hypotension | 1 hour after dialysis start during a single session.
  PFVV represents the variation in peak flow velocity in the carotid artery measured by ultrasonography at 1 hour after hemodialysis start. It reflects vascular volume status and elastic properties. Its capacity to predict intradialytic hypotension will be assessed through sensitivity, specificity, and ROC analysis.

SECONDARY OUTCOMES:
Incidence of Intradialytic Hypotension | Up to 1 dialysis session (4 hours)
  The proportion of dialysis sessions in which patients experience hypotension, defined as a decrease in systolic blood pressure (SBP) of 20 mmHg or more during the session, will be recorded to estimate clinical event frequency.
Correlation Between FTc and PFVV and Changes in Blood Pressure | 1 hour after dialysis start during a single hemodialysis session (total duration up to 4 hours)
  Assessment of the statistical correlation between PVI parameters ( FTc and PFVV) and changes in blood pressure, including systolic blood pressure, diastolic blood pressure, and mean arterial pressure, during the dialysis session.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Wannan Medical College (Yijishan Hospital of Wannan Medical College), Wuhu, Outside of the US, China

IPD SHARING:
Plan to Share IPD: No